CLINICAL TRIAL: NCT06308029
Title: Effectiveness of an eHealth Self-management Support Program for Persistent Pain After Breast Cancer Treatment
Acronym: PECAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); University Ghent (Other); KU Leuven (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, An De Groef, Assistant Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Edge003203; T001122N (Other Grant/Funding Number: Research Foundations Flanders); s68058 (Other: UZ/KU Leuven ID)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: eHealth; pain; active lifestyle; pain management; physiotherapy
MeSH Terms: conditions — Breast Neoplasms; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized, multi-centric, three-arm controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- eHealth self-management support program (Experimental): This web-based eHealth program consists of two parts. First participants will complete a pain science education program. After being primed in the educational program, barriers for a physically active lifestyle should be removed and participants should be able to apply the learned information in the second part. The second part of the self-management support program consists of daily activity planning and strategies to promote an active lifestyle.
  Interventions: Behavioral: eHealth self-management support program
- Face-to-face rehabilitation program (Active Comparator): The face-to-face rehabilitation program combines pain science education with an active behavioral approach. First, 2-3 individual face-to-face sessions are organized with a physical therapist (recruited and trained by the research team) to provide pain science education. The content of this pain science education program is the same as for the eHealth program. Similar as in the eHealth program, this education intervention includes advice for activity management, while experiencing pain and other symptoms, in order to remove barriers for an active lifestyle. The educational information will be presented verbally (explanation by the therapist) and written (information leaflet, summaries, pictures, metaphors and diagrams on computer and paper). After the education, the physical therapist will discuss proper goal setting with the patient to reach an active lifestyle and will coach the participant to reach these goals with maximum 6 face-to-face sessions.
  Interventions: Behavioral: Face-to-face rehabilitation program
- Usual care group (No Intervention): Usual care for breast cancer survivors with persistent pain consists of primarily a pharmacological approach and general advice to stay or become active. This information is given to the participant by means of a brochure.

INTERVENTIONS:
Behavioral: eHealth self-management support program — This web-based eHealth program consists of two parts. First participants will complete a pain science education program. After being primed in the educational program, barriers for a physically active lifestyle should be removed and participants should be able to apply the learned information in the second part. The second part of the self-management support program consists of daily activity planning and strategies to promote an active lifestyle. The eHealth program will be accessible from any digital device (laptop, tablet, smartphone) after receiving a personal login code provided by the researcher. Participants go through the eHealth program independently at their own pace. It is recommended to do this in 8-12 weeks.
  Arms: eHealth self-management support program
Behavioral: Face-to-face rehabilitation program — The face-to-face rehabilitation program combines pain science education with an active behavioral approach. First, 2-3 individual face-to-face sessions are organized with a physical therapist to provide pain science education. The content of this pain science education program is the same as for the eHealth program. Similar as in the eHealth program, this education intervention includes advice for activity management, while experiencing pain and other symptoms, in order to remove barriers for an active lifestyle. The educational information will be presented verbally and written. After the education, the physical therapist will discuss proper goal setting with the patient to reach an active lifestyle and will coach the participant to reach these goals with maximum 6 face-to-face sessions. It is recommend to organise the in total 9 face-to-face sessions within a periode of 8-12 weeks.
  Arms: Face-to-face rehabilitation program

SUMMARY:
The scientific goals of the project are:

1. The primary scientific objective of the study is to determine the effectiveness of an eHealth self-management support program for persistent pain after breast cancer treatment compared to:

   * usual care (i.e. superiority of the eHealth self-management support program) and
   * a comprehensive pain rehabilitation program delivered face-to-face in a physical therapy setting (i.e. non-inferiority of the eHealth self-management support program)

   on pain-related disability (measured with the Pain Disability Index).
2. The secondary scientific objectives of this study entails to examine if the eHealth self-management support program has a relative benefit for other biopsychosocial factors, including:

   * Other dimensions of pain
   * Health-related quality of life
   * Physical functioning, including physical activity levels
   * Psychosocial functioning, including self-efficacy, stress, anxiety, depression, coping style (key secondary outcome) and fear of cancer recurrence
   * Participation in society, including return to work
   * Healthcare-related costs for the patient and society
3. The tertiary scientific objectives of this study are

   * to identify moderators of treatment effect, including behavioural determinants (e.g. self-efficacy, motivation, coping style), in order to identify breast cancer survivors who would benefit the most of the eHealth self-management support program and to allow more stratified and efficient pain management care and more targeted allocation of budgets.
   * To examine the implementation process, mechanisms of impact and contextual factors.

DETAILED DESCRIPTION:
The current state-of-the art advocates for a biopsychosocial rehabilitation approach for persistent pain after breast cancer treatment. Within this approach pain science education is combined with promotion of an active lifestyle based on self-regulation techniques. The investigators argue for testing an innovative eHealth self-management support program for this purpose. The assumption is that this delivery mode reduces barriers to pain self-management support, by bringing timely support near to people, creating a safe environment as opposed to hospital settings, providing a multidimensional support model taking into account the biopsychosocial needs of patients, and lowering costs. This program can provide patients with the knowledge, proactive, cognitive and self-management skills to master their situation and journey towards less pain and pain-related disability and participation in normal life again. Therefore, the general aim of the proposed project is to investigate the effectiveness of an eHealth self-management support program for pain-related disability (I) in breast cancer survivors with persistent pain (P). The program makes use of an innovative chatbot format for delivering pain science education and motivating and monitoring physical activity. The eHealth program is automated using comprehensive decision-tree-based algorithms in order to promote pain self-management support. The primary scientific objective of the study is to determine the effectiveness of this eHealth self-management support program for persistent pain after breast cancer treatment compared to 1) usual care (i.e. superiority of the eHealth self-management support program) (C1) and 2) a comprehensive pain rehabilitation program delivered face-to-face in a physical therapy setting (i.e. non-inferiority of the eHealth self-management support program) (C2) on pain-related disability (O).

ELIGIBILITY:
Inclusion criteria

* Patients (men and women) with primary breast cancer and with unilateral or bilateral axillary surgery (Axillary Lymph Node Dissection or Sentinel Node Biopsy);
* Be non-metastatic and have finished their primary treatment with a curative intent at least 3 months prior to study participation;
* Adjuvant hormonal therapy and immunotherapy form the exception to the rule are tolerated;
* Presence of self-reported persistent pain in the last 3 months that interferes with daily activities (yes/no)

Exclusion criteria

* Can not participate during the entire study period;
* Mentally or physically unable to participate in the study;
* Previous participation in a pain science education program.
* No acces to a digital device
* Do not speak/understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pain-related disability | at 6 months follow-up
  Measured with Pain Disability Index, an instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. Scores between 0 and 70. The higher the score the greater the person's disability due to pain. The trial will be termed successful when superiority of the eHealth self-management to usual care and non-inferiority of the eHealth self-management program to face-to face rehabilitation program has been shown for the primary outcome at 6 months. Both tests will be based on the comparison of the mean value after correction for the baseline PDI (ANCOVA approach).

SECONDARY OUTCOMES:
Pain related disability | at 12 weeks and 12 months follow-up
  Measured with Pain Disability Index, an instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. Scores between 0 and 70. The higher the score the greater the person's disability due to pain
Pain severity | at 12 weeks, 6 months and 12 months follow-up
  Measured with a Visual Analogue Scale (0-100), a higher score indicates more severe pain.
Severity of neuropathic Pain | at 12 weeks, 6 months and 12 months follow-up
  Measured with the Neuropathic Pain Symptom Inventory (0-100), a higher score indicates more severe pain.
Medication use | at 12 weeks, 6 months and 12 months follow-up
  self-composed questionnaire
Pain location | at 12 weeks, 6 months and 12 months follow-up
  Margolis Pain Diagram
Knowledge of neurophysiology of pain | at 6 weeks
  measured with the Neurophysiology of Pain Test
Physical Activity pattern | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patterns of Activity Measure - Pain (short form). It measures 3 pain-related activity patterns: avoidance, overdoing, and pacing. Potential scores on each of the 3 POAM-P scales can range from 0 to 20. Higher scores in any pattern indicate more of the measured construct.
Physical functioning | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Fatigue | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System( PROMIS)-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Sleep disturbance | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Pain Beliefs | at 6 weeks, 12 weeks, 6 months and 12 months follow-up
  Measured with the Survey of Pain Attitudes (SOPA)-short form. It contains seven subscales including 30 items in total with a 5-item Likert scale. Each domain of the SOPA is expressed as a score compared to the average of a group (T-score).
Pain-related worrying | at 12 weeks, 6 months and 12 months follow-up
  Measured with the Pain Catastrophizing Scale. Thirteen items are scored on a 5-item Likert scale ranging from "not" to "always". The total score ranges from 0 to 52, where higher scores are associated with higher levels of catastrophizing.
Vigilance and interpretation of physical sensations | at 12 weeks, 6 months and 12 months follow-up
  Measured with the Bodily Threat Monitoring Scale. This is a new 19-item self-report measure that captures the tendency to monitor and interpret bodily sensations as symptomatic of something being wrong with one's body. Scores range from 0 to 76, with higher scores indicating greater bodily threat monitoring.
Depression | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 Profile v2.01.Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Anxiety | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Determinants for physical activity | at 12 weeks, 6 months and 12 months follow-up
  measured with the Determinants of Physical Activity Questionnaire. Each item was assessed using a 7-point scale for all determinants of physical activity. Lower scores indicate low exercisers, while high scores indicate high exercisers.
Participation | at 12 weeks, 6 months and 12 months follow-up
  measured with the PROMIS-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Well-being | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health. Each domain of the PROMIS is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Social Support | at 12 weeks, 6 months and 12 months follow-up
  measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 Profile v2.01. Each domain of the PROMIS-57 is expressed as a score compared to the average of a group (T-score). A T-score is a standardized score. The average score in a population is assigned the value 50. The standard deviation becomes equated to 10 points.
Return to work rate | at 12 weeks, 6 months and 12 months follow-up
  measured with a self-composed questionnaire
Medical costs of medical consumption | at 12 weeks, 6 months and 12 months follow-up
  measured with the Medical Consumption Questionnaire. The costs of medical consumption are calculated by measuring the volumes of care multiplied by the cost price per unit of care.
Indirect costs related to disease outside health care | at 12 weeks, 6 months and 12 months follow-up
  measured with the Productivity Cost Questionnaire. To calculate the costs of production losses, volumes are multiplied with unit costs.
Health-related quality of life | at 12 weeks, 6 months and 12 months follow-up
  measured with the EuroQol-5Dimensions-5Levels (EQ-5D-5L) questionnaire. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Standard EQ-5D-5L value sets are available for different regions. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Patient Global Impression of Change | at 12 weeks follow-up
  measured with the Patient Global Impression of Change (PGIC). PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: An De Groef, PhD, Principal Investigator — Universiteit Antwerpen; Nele Devoogdt, PhD, Principal Investigator — KU Leuven; Geert Crombez, PhD, Principal Investigator — UGent
Locations (2):
- Belgium (2):
  - Universiteit Antwerpen, Antwerp
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Yes
The data are not openly available and are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: on request
Access Criteria: on request

REFERENCES:
- [Derived] De Groef A, Dams L, Moseley GL, Heathcote LC, Wiles LK, Catley M, Vogelzang A, Hibbert P, Morlion B, Van Overbeke M, Tack E, Van Dijck S, Devoogdt N, Gursen C, De Paepe AL, Mertens M, van Olmen J, Willem L, Tjalma W, Nevelsteen I, Neven P, Vanhoudt R, Wildemeersch D, De Backere F, Fieuws S, Crombez G, Meeus M. Study protocol for a pragmatic randomised controlled trial in Belgian primary care and hospital settings on the effectiveness of an eHealth self-management support programme consisting of pain education and coaching of activity needs in breast cancer survivors with persistent pain: the PECAN trial. BMJ Open. 2025 Aug 22;15(8):e099241. doi: 10.1136/bmjopen-2025-099241. PMID 40846340